CLINICAL TRIAL: NCT03161769
Title: MAX-PIPE Registry - Maximizing Flow Diversion Effect On The Treatment of Large Intracranial Aneurysms With PIPEline Flex Embolization Devices Using Optical Flow Imaging Software "AneurysmFlow"
Brief Title: MAXimizing Flow Diversion Effect On the Treatment of Large Intracranial Aneurysms With Embolization Devices
Acronym: MAX-PIPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Vitor Pereira, Associate Professor of Radiology and Surgery, University Health Network, Toronto
Other Study IDs: TWH -Version 4.0 July 13 2016
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Percutaneous neurovascular treatment: Procedure: Percutaneous neurovascular treatment of intracranial aneurysms
  Interventions: Procedure: Neurovascular treatment of intracranial aneurysms; Device: AneurysmFlow image processing software

INTERVENTIONS:
Procedure: Neurovascular treatment of intracranial aneurysms — Endovascular treatment of intracranial aneurysms using flow diverting stents
Device: AneurysmFlow image processing software — Software to process and display images of intracranial aneurysm treatment using flow diverting stents.

SUMMARY:
Investigate the ability of the intra-operative, intra-aneurysmal flow evaluation to assist with the treatment of intracranial large aneurysms using Embolization Device(s)

DETAILED DESCRIPTION:
The Division of Neuroradiology at UHN (Toronto Western Hospital) would like to initiate a single center registry study on the treatment of large intracranial aneurysms with PIPEline[tm] flex embolization devices using optical flow imaging software, "AneurysmFlow". The study team will consent patients diagnosed with unruptured brain / intracratial aneurysms IA(s) . The selected patients ,who booked for elective brain aneurysm repair/endovascular treatment with Flow diverter devices (FDS) called Pipeline embolization devices (PED), will qualify for registry participation . During the PED procedure, the study team will be using AneurysmFlow software to calculate a new metric called the MAFA ratio (Mean Aneurysm Flow Amplitude). By calculating the MAFA ratios intra-operatively, the interventionalist can adapt the therapeutic strategy in order to maximize the flow diverting effect on inducing complete aneurysm occlusions (thrombosis). Additionally, the purpose of this study is to further expand the body of clinical knowledge concerning the relationship between blood flow metrics as determined by the AneurysmFlow software and clinical outcome in patients undergoing treatment for intracranial aneurysms (IAs) with Pipeline and Pipeline Flex embolization devices. The study team aims to collect data at a 12 month follow-up period for each patient

ELIGIBILITY:
Inclusion Criteria:

1. Subject with unruptured, large (≥8mm) saccular aneurysm(s) located in the anterior intracranial circulation and suitable for an endovascular treatment with a Flow Diverter Stent.
2. Subject has signed an institutionally approved research informed consent form.
3. Subject ≥ 18 years old.

Exclusion Criteria:

1. Subject with non-saccular brain aneurysm (s) such as:- dissecting; fusiform; atherosclerotic; mycotic; bifurcational.
2. Subject underwent a prior target brain aneurysm treatment with either endovascular (stenting, coiling) or surgical (clipping) techniques.
3. The endovascular treatment of subject's target aneurysm(s) was assisted with coils or intracranial stents (non-FDS) before the AneurysmFlow calculations.
4. Subject with partially thrombosed or recanalized target brain aneurysm(s).
5. Subject had prior significant or severe allergy to intra-arterial contrast medium uncontrolled by pre-procedure medications.
6. Subject with severe kidney disease (e-GFR < 60).
7. Subject is not willing (or not able) to attend post FDS insertion follow up clinic visits requiring DSA, head MRI or CTA imaging.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with unruptured saccular Intracranial Aneurysms IA(s) suitable for endovascular treatment with PIPEline™ Embolization Devices or PIPEline™ Flex Embolization Devices.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-04-21 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete aneurysm occlusion at 12 months based on contrast agent volume measurement in angiography. | 1 year
  ≥86% complete aneurysm occlusion rate after 12 months post-treatment using optical flow analysis with a MAFA threshold ratio of 0.89, measured with an image processing tool.

SECONDARY OUTCOMES:
Number of participants with complete aneurysm occlusion at 6 months based on contrast agent volume measurement in angiography. | 6 months
  ≥74% complete aneurysm occlusion rate after 6 months post-treatment using optical flow analysis with a MAFA threshold ratio of 0.89, measured with an image processing tool.
High sensitivity and specificity (> 80%) of the MAFA ratio to determine aneurysm occlusion rates based on ROC statistical calculations. | 1 year
  Data collected from the registry will be used to help determine a new, more optimal MAFA ratio threshold for predicting post-FDS aneurysm occlusion at 12 months post-treatment based on receiver operating characteristic (ROC) statistical curves.
Number of participants with treatment complications as assessed by an electronic patient record. | 1 year
  Predictability of the MAFA ratio for treatment complications (aneurysm rupture, in-stent thrombosis, mass effect, using a correlation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Vitor Pereira, MD, Principal Investigator — Associate Professor or Radiology and Surgery
Locations (1):
- Toronto Western Hospital - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No